CLINICAL TRIAL: NCT01991834
Title: Antibiotic Prophylaxis in Gynecologic Laparoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Fabiola Soares Moreira Campos, MD, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MPFabiola
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Infection Secondary to Surgical Procedure
Keywords: laparoscopy; surgical wound infection; antibiotic prophylaxis; gynecologic surgical procedures
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cefazolin; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Patients in this arm will receive intravenous sterile saline 30 minutes before the gynecologic laparoscopy.
  Interventions: Procedure: gynecologic laparoscopy; Drug: Placebo
- Cefazolin (Active Comparator): Patients in this arm will receive intravenous cephazolin 1g, 30 minutes before the gynecologic laparoscopy.
  Interventions: Procedure: gynecologic laparoscopy; Drug: Cefazolin

INTERVENTIONS:
Procedure: gynecologic laparoscopy — Gynecological laparoscopy without opening hollow viscera.
  Other Names: pelvic laparoscopy; gynecologic laparoscopic surgery
Drug: Cefazolin — Intravenous administration of 1 g of cefazolin
  Other Names: Cephazolin; Cefazoline; Cephazolin Sodium for Injection; Kefzol
  Arms: Cefazolin
Drug: Placebo — Intravenous administration of saline sterile solution
  Other Names: placebo treatment
  Arms: Placebo

SUMMARY:
Laparoscopy is a surgical procedure indicated for most gynecological pathologies and presents numerous advantages over laparotomy, among them lower rates of surgical site infection and less comorbidity feverish. Despite this, the use of antibiotic prophylaxis is widely accepted and performed by most gynecologists. However, there isn't literature evidence to support the routine use of antibiotics in the prophylaxis of wound infection on laparoscopic pelvic surgery .Therefore, this study will evaluate the need for the use of antibiotic prophylaxis in gynecological laparoscopies not including opening hollow viscera.

DETAILED DESCRIPTION:
It is a clinical, prospective, double-blind, randomized study. 114 women with gynecologic disease, in which there is indication of laparoscopic surgical approach, will be consecutively select. These women will be allocated in two arms, control and study, where control group will use placebo and study will receive intravenous cephazolin. These patients will be followed for 30 days according to Centers for Disease Control and Prevention criteria.

ELIGIBILITY:
Inclusion Criteria:

* patients with gynecologic disease, undergoing gynecologic laparoscopy without opening hollow viscera.

Exclusion Criteria:

* body mass index over 30 Kg/m2
* smoking
* diabetes type I or II with glycated hemoglobin exceeding 6.5%
* patients who are at surgical risk classification of the American Society of Anesthesiologists(ASA) as ASA III or higher
* refusal to participate
* postoperative antibiotic therapy for another indication clinical complication

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-09; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 30 days
  Patients are followed weekly by a masked surgeon in regard to surgical site infecton (SSI), until the 30th postoperative day. Centers for Disease Control and Prevention's (CDC) criteria and classification were adopted.

CONTACTS AND LOCATIONS:
Overall Officials: Fabiola SM Campos, MD, Principal Investigator — Universidade do Vale do Sapucai; Daniela F Veiga, MD, PhD, Study Chair — Universidade do Vale do Sapucai
Locations (2):
- Brazil (2):
  - Hospital das Clinicas Samuel Libanio, Pouso Alegre, Minas Gerais
  - Hospital e Maternidade Santa Paula, Pouso Alegre, Minas Gerais